CLINICAL TRIAL: NCT00765700
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 3 Study to Assess the Efficacy and Safety of Ketotransdel™ (Ketoprofen Topical Cream 10%) in the Treatment of Pain Associated With Mild to Moderate Acute Soft Tissue Injury.
Brief Title: Ketoprofen 10% Cream for Treatment of Pain Associated With Mild to Moderate Acute Soft Tissue Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imprimis Pharmaceuticals, Inc. (Industry)
Collaborators: Cato Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDLP-110-101
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Sprain; Strain; Acute Soft Tissue Injury
Keywords: Sprain; Strain; Pain; Ankle Pain; Shoulder Pain; Elbow Pain; Tennis Elbow; Knee pain; Wrist Pain; Hand Pain; Muscle, Bone and Cartilage Disorders
MeSH Terms: conditions — Sprains and Strains; Pain; Shoulder Pain; Tennis Elbow; Cartilage Diseases | interventions — Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketoprofen 10% Cream (Active Comparator): Topical Ketoprofen 10% Cream
  1gram three times daily for 7 days
  Interventions: Drug: Topical Ketoprofen 10% Cream
- Placebo (Placebo Comparator): Topical placebo cream
  1gram three times daily for 7 days
  Interventions: Drug: Topical Placebo Cream

INTERVENTIONS:
Drug: Topical Ketoprofen 10% Cream — Topical Administration
  Other Names: Ketotransdel (TDLP-110)
  Arms: Ketoprofen 10% Cream
Drug: Topical Placebo Cream — Topical Administration
  Other Names: Placebo; Vehicle
  Arms: Placebo

SUMMARY:
Imprimis Pharmaceuticals is investigating a proprietary, topical cream formulation consisting of 10% ketoprofen (containing 100 mg of ketoprofen in 1gram of cream) for the local treatment of acute musculoskeletal pain.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the efficacy and safety of ketoprofen 10% cream compared to placebo as a three-times-per-day topical application in improving the patient assessment of pain when used to treat mild to moderate acute soft tissue injury of the upper and lower extremities over a 7-day period.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age
* Have a diagnosis of uncomplicated acute soft tissue injury of the upper or lower extremity that has occurred within the 72 hours preceding the baseline visit.
* The injury site must be accessible to the patient so that he or she can apply the study treatment himself or herself.
* Meet pain entry criteria.
* Willing to discontinue use of any pain medication or treatments not provided as part of the study.

Exclusion Criteria:

* Grade 3 sprain or strain, bilateral sprain or strain, or concomitant fracture or open wound at the site of the sprain or strain, or have a serious injury, as determined by the investigator (e.g., nerve damage, joint instability, or tendon rupture).
* Previous injury to the same area within 3 months prior to current injury.
* Active skin lesions or disease at the intended site of application of the study medication. Skin lesions include open wounds, rash, papules, vesicles, and erythema associated with the site of injury.
* Pharmacologic treatment (NSAIDs or analgesic medications) for the injury less than 12 hours before the baseline assessments.
* Any form of opioid use since the time of injury.
* Any form of steroid use within 30 days prior to study entry.
* Non-pharmacologic treatments of the injury other than rest, ice, compression, and/or elevation (RICE) prior to the baseline visit.
* History or physical examination finding that is not compatible with safe participation in the study as determined by the study doctor, such as gastrointestinal (stomach, intestine) ulcer or bleeding within 6 months documented by an upper-gastrointestinal series (UGI x-ray, barium meal) or endoscopy (GI scope), anemia or abnormal bleeding, moderate to severe kidney disease, or moderate to severe liver disease.
* A history of, or evidence for, underlying disease in the injured area, such as osteoarthritis or gout.
* Clinically significant, poorly controlled lung, stomach, liver, kidney, heart, or other vital organ disease as determined by the study doctor or nurse.
* A history of allergy to ketoprofen or ketoprofen-containing products.
* A history of allergy to soy lecithin or soy lecithin-containing products.
* Medications (drugs) or other substances contraindicated due to the nature of study medication that include:

  * Allergies to prescription or over-the-counter products containing acetaminophen (e.g., Tylenol®), which is used as rescue medication
  * History of aspirin-sensitive asthma, or aspirin-associated rhinitis or nasal polyps
  * Taking warfarin, parenteral heparin, ticlopidine or clopidogrel
  * Taking lithium or methotrexate
  * Taking probenecid or similar drugs that might affect the kidneys
* Received an investigational drug or product or participated in an investigational drug study within a period of 30 days prior to receiving study medication.
* Scheduled elective surgery or other invasive procedures during the period of study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of ketoprofen 10% cream in subjects with acute pain associated with mild to moderate acute soft tissue injury (acute sprain or strain) of upper and lower extremities on the day 3 visit. | 7 days

SECONDARY OUTCOMES:
Assess the safety, tolerability and other parameters of ketoprofen 10% cream in subjects with acute pain associated with mild to moderate acute soft tissue injury of upper and lower extremities. | 14 days

OTHER OUTCOMES:
To assess the pharmacokinetics of ketoprofen after 7 days of topical application | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Illana Katsnelson, MD, Study Director — Cato Research
Locations (1):
- CATO Research, Durham, North Carolina, United States

REFERENCES:
- [Result] E. Ekman, S. Skrepnik, M. Jones , K. Lawson, and J. Schupp. EFFICACY AND SAFETY OF KETOPROFEN 10% CREAM IN ACUTE SOFT TISSUE INJURIES (PHASE 3 STUDY TDLP-110-001). Poster Presentation, Sep. 2, 2010, 13th World Congress on Pain in Montreal, Canada.